CLINICAL TRIAL: NCT07082998
Title: Comparing the Efficacy of Heated Yoga and Sauna as a Treatment for Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Maren Nyer, clinical psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025P001188
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Depression Disorders; Depression - Major Depressive Disorder; Depression Disorder; Depression Chronic; Depression; Depression in Adults
Keywords: depression; heated yoga; yoga; sauna; mindfulness; mindfulness app; clinical trial
MeSH Terms: conditions — Depression | interventions — Steam Bath

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- heated yoga (Experimental): heated yoga 2x per week for 12 weeks
  Interventions: Behavioral: heated yoga
- sauna (Experimental): infrared sauna 2x per week for 12 weeks
  Interventions: Behavioral: sauna
- mindfulness app (Active Comparator): Insight Timer app for 80 mins per week for 12 weeks
  Interventions: Behavioral: mindfulness app

INTERVENTIONS:
Behavioral: heated yoga — 12-weeks of twice weekly 90-min heated yoga classes in the community
  Arms: heated yoga
Behavioral: sauna — 12-weeks of twice weekly 40-min sauna sessions in the community
  Arms: sauna
Behavioral: mindfulness app — 12-weeks of 80-mins a week of a mindfulness app
  Arms: mindfulness app

SUMMARY:
This project explores whether heated yoga, sauna, and a mindfulness app reduce depressive symptoms

DETAILED DESCRIPTION:
This is a parallel group study design. The investigators plan to enroll 120 adults who have at least moderate depression and will be randomized in an equal allocation ratio (i.e., 1:1:1) across three groups: heated yoga vs. sauna vs. a mindfulness app. The interventions will be provided over a 12-week period and assessments will occur at baseline (Week 0), mid-intervention (Weeks 4 & 8), post-intervention (Week 12, primary outcome), and at a 4-week (Week 16). Then participants enter an optional 1-month choice intervention period with a post-assessment (Week 20).

ELIGIBILITY:
Subject Characteristics

Inclusion Criteria:

1. adults (18-65 years old)
2. Ability to provide informed consent
3. English language proficiency
4. PHQ-9 score > 10, indicating at least moderate depressive symptoms 21
5. Must have filled out the waiver for the community-based partners prior to enrolling in the study*
6. Individuals of childbearing potential must use an acceptable form of birth control
7. (if applicable) willingness to keep psychiatric medications and psychotherapy stable throughout the course of the study
8. Must be able to access mindfulness app on a device (i.e., smartphone, iPad, etc.)
9. Can travel to Breathe in Harvard Square and at least one Restore location (i.e., Hingham, Somerville, Dedham, Newton, Lynnfield)

Exclusion Criteria:

1. Pregnant or planning to become pregnant
2. Breast feeding
3. Active suicidal thinking (i.e., PHQ-9 item 9 ≥1 and a positive response to C-SSRS screener items 3, 4, 5, or 6)
4. Active eating disorders or substance use disorders within the past 12 months, as per the MINI
5. Primary OCD or PTSD, as per the MINI
6. History of bipolar disorder, psychotic disorders, as per the MINI
7. ≥25% drop in PHQ-9 score from screen to baseline
8. Under the influence or withdrawal of drugs or alcohol
9. Positive urine toxicology screen due to illicit drug use or other exclusionary medications. (Potential false positives will be addressed on a case-by-case basis at the discretion of the PI or designee)
10. have had a bone fracture or joint surgery in the past 6 months
11. not able to walk freely or without difficulty
12. any serious, unstable medical condition as determined by the revised Physical Activity Readiness Questionnaire (PAR-Q+) and do not have approval from their treating physician (we will check in with treating physician in the event that participants endorse any item on the PAR-Q+)
13. participants must have a healthcare provider who they could contact if they needed medical care, such as a primary care doctor, a counselor, a psychiatrist, a nurse practitioner, or a clinic that you go to.
14. Significant exposure to heated yoga classes in the past 3 months (i.e., more than 6 classes)
15. Significant exposure to sauna sessions in the past 3 months (i.e., more than 6 sessions)
16. Significant exposure to mindfulness app in the past 3 months (i.e., more than 6 uses of the app)
17. are on medications that make dehydration more likely (e.g., lithium, antipsychotics, insulin-dependent) diuretics, barbiturates, b-blockers, anticholinergics, current ETOH acute intoxication, reduced ability to sweat, hemophilia, pacemaker (magnets used to assemble saunas can interrupt the pacer)
18. antidepressant or psychiatric medications that are initiated less than 8 weeks or a dose change less than 4 weeks prior to screening visit
19. psychotherapy that has been initiated within the past 3 months
20. psychiatric hospitalization within the past year
21. diagnosed with any neurological disorders that would impact participation or make participation unsafe
22. are currently in active ketamine, Electroconvulsive therapy, or Transcranial Magnetic Stimulation treatments
23. are unable to follow the study procedures (e.g., not able to travel to the heated yoga or sauna studios)
24. A subject who in the opinion of the Principal Investigator would not be able to safely complete the study or would jeopardize study integrity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Weeks 0, 4, 8, 12, 26, 20
  The PHQ- 9 is a 9-item self-report questionnaire that is widely used to assess depression symptom severity. Score range from 0 to 27, with a high score (20-27) indicating severe depression.

SECONDARY OUTCOMES:
The Five Facet Mindfulness Questionnaire (FFMQ-15) | Weeks 0, 4, 8, 12, 16, 20
  A 15-item self-report instrument that measures mindfulness; derived from factor analytic study of five independent mindfulness questionnaires. Total scores range from 15 to 75, with higher scores indicating greater utilization of mindfulness techniques.
Ruminative Responses Scale (RRS) | Weeks 0, 4, 8, 12, 16, 20
  A 22-item questionnaire that assess rumination, with scores range from 22 to 88. Lower scores reflect less frequent engagement in ruminative thought patterns.
The World Health Organization-5 Well-Being Index (WHO-5) | Weeks 0, 4, 8, 12, 16, 20
  A 5-item self-report questionnaire with positively-worded statements related to general mood over the prior two weeks. WHO-5 has shown strong construct validity as a measure of general quality of life, and is sensitive to change. Scores range from 0 to 25, with higher scores reflecting overall well-being.
Patient-Reported Outcomes Measurement Information System (PROMIS-29) | Weeks 0, 4, 8, 12, 16, 20
  PROMIS-29 is used to assess psychometric properties under the domains of physical function, fatigue, pain interference, depressive symptoms, anxiety, social functioning, sleep disturbance using four items per domain. This measure uses a T-score metric for scoring, typically ranging from 20 to 80, with a lower T-score (below 50) indicating less severity of symptoms.

OTHER OUTCOMES:
Acceptability Interview | Week 12
  Used to evaluate participants' thoughts about the study and collect information on their experience. The data collected is qualitative.

CONTACTS AND LOCATIONS:
Overall Officials: Maren B Nyer, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No